CLINICAL TRIAL: NCT00777361
Title: An Open, Two Period, Single Dose, Phase I Study of the Excretion of Radioactivity, Metabolic Profiles and Pharmacokinetics Following Oral Administration of [14C]-AZD3480 and the Pharmacokinetics of AZD3480 Following Intravenous Administration to Healthy Male Volunteers With Different CYP2D6 Genotype
Brief Title: Study of Uptake, Break Down and Elimination of an Investigational Drug in Healthy Volunteers
Acronym: MB
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn Paulsson, MD, PhD, Medical Science Director Clinical Neuroscience TA, AstraZeneca R&D Södertälje
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D3690C00017; EudraCT No.: 2007-005903-16
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer's Disease
Keywords: Mass balance; AZD3480, Pharmacokinetics, Healthy volunteers
MeSH Terms: conditions — Alzheimer Disease | interventions — ispronicline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AZD3480 iv (Experimental): Single iv infusion AZD3480
  Interventions: Drug: AZD3480
- Oral [14C] AZD3480 (Experimental): Single oral dose [14C]AZD3480
  Interventions: Drug: AZD3480

INTERVENTIONS:
Drug: AZD3480 — Iv single dose, 4-hour infusion of 25 mg
  Arms: AZD3480 iv
Drug: AZD3480 — Oral solution single dose of 50 mg
  Arms: Oral [14C] AZD3480

SUMMARY:
This study is being performed in order to learn more about a new drug (possible as treatment for people with Alzheimer's Disease and other conditions with cognitive dysfunction (memory and attention problems)) and how it is handled by the body by giving the drug to healthy volunteers with different genotypes.

ELIGIBILITY:
Inclusion Criteria:

* Physically healthy volunteers
* Participation in a previous study for genotyping for identification to be extensive, intermediate or poor metaboliser (CYP2D6 enzyme)

Exclusion Criteria:

* History of clinically significant diseases or illness.
* Ues of any prescribed or non-prescribed medications from 2 weeks prior to first treatment day except for paracetamol and OTC adrenergic nasal spray.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Recovery (% dose) of radioactivity retrieved in urine and faeces Total radioactivity in blood and plasma, AUC, Cmax , tmax, t1/2 and blood/plasma ratio. | Urine and faeces collection for at least 168 hours (up to 2 weeks)9 (blood) and 17 (plasma) samples during 48 and 72 hours.
Plasma and urine concentration (AUC, Cmax, tmax, t1/2, F, CL, CLR, fe, Ae, and Vss) | 19 and 18 blood samples during 72 and 96 hours after iv (Visit 2) and po dosing (Visit 3) respectively. Urine collection for 72 hours and 168 hours (up to 2 weeks).

SECONDARY OUTCOMES:
identity of major metabolites in plasma and excreta | 4 blood samples during 8 hours.Urine and faeces collection for at least 168 hours (up to 2 weeks).
Adverse Events, vital signs (supine blood pressure and pulse rate), ECG, hematology, clinical chemistry and urinalysis. | From enrollment to follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Björn Paulsson, MD, PhD, Study Director — AstraZeneca Södertälje, Sweden; Tim Mant, Prof, Principal Investigator — Quintiles Drug Research Unit @ Guy´s Hospital
Locations (1):
- Research site, Macclesfield, Cheshire, United Kingdom